CLINICAL TRIAL: NCT06334042
Title: Examination of the Effects of Chromium Levels on Glucose Metabolism, Lipid Metabolism, Morbidity and Mortality Rates in Patients Followed in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Oguzhan Kahveci (Other)
Responsible Party: Sponsor-Investigator, Oguzhan Kahveci, Anesthesiology Resident, MD, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: GO 23/488
Record Dates: First submitted 2024-03-12; First posted 2024-03-27 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Chromium Deficiency; Diabetes Mellitus; Hyperlipidemias; Hypercholesterolemia
Keywords: Intensive care; Metabolism,glucose; Metabolism,lipid
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive Care Patients
  Interventions: Diagnostic Test: Serum Chromium Level

INTERVENTIONS:
Diagnostic Test: Serum Chromium Level — Measuring serum chromium levels from patients who admitted in intensive care unit.

SUMMARY:
The goal of this observational study is to determine the effects of chromium serum levels on glucose metabolism, lipid metabolism, morbidity and mortality rates in critically ill intensive care patients. The investigators' goal is to provide a different perspective on solving the common problems of hyperglycemia and dyslipidemia encountered in intensive care patients, aiming to reduce morbidity and mortality rates.

Participants will give a single blood sample (into trace element serum sample tube) on the day of admission to the intensive care unit, along with routine blood tests, and samples will be taken once a week during their stay in the intensive care unit.

DETAILED DESCRIPTION:
Hyperglycemia is a common risk factor in critically ill patients admitted to intensive care units; increasing hospital stay duration, morbidity/mortality rates and is associated with increased undesirable cardiovascular events, thrombosis, inflammatory changes, impaired immune functions, increased infection frequency, delayed wound healing, osmotic diuresis, fluid - electrolyte imbalances and other issues.

Dyslipidemia plays a significant role in the development of atherosclerosis and consequently cardiovascular disease.

Chromium (Cr) is a trace metal. It has been claimed that trivalent chromium is a cofactor of a low molecular weight chromium - binding substance (LMWCr; also known as chromodulin), an oligopeptide. LMWCr can enhance the action of insulin, thereby improving tissue insulin sensitivity and facilitating glucose transport into the cells. This hypothesis is supported by observations that chromium deficiency leads to an increase in blood sugar, total cholesterol and triglycerides; a decrease in high - density lipoproteins (HDL) and insulin sensitivity.

Patients aged 18 and older admitted to the Intensive Care Unit of Hacettepe University Department of Anesthesiology will be included in the study. A single blood sample (into trace element serum sample tube) will be taken from participants in the study group on the day of admission to the intensive care unit, along with routine blood tests, and samples will be taken once a week during their stay in the intensive care unit. The chromium level in the collected blood samples will be analyzed using inductively coupled plasma - mass spectrometry (ICP - MS). The laboratory results of the monitored participants will be prospectively recorded in the data collection form and in International Business Machines Statistical Product and Service Solutions (IBM SPSS).

A literature review revealed very few publications on the effects of chromium serum levels on glucose metabolism, lipid metabolism, morbidity and mortality rates; and the existing publications did not include samples of critically ill intensive care patients. With this study, the investigators aim to contribute to the national and international literature with a large sample of intensive care patients. Thus, the investigators' goal is to provide a different perspective on solving the common problems of hyperglycemia and dyslipidemia encountered in intensive care patients, aiming to reduce morbidity and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Admitted to Anesthesiology Intensive Care Unit

Exclusion Criteria:

* Patient Refusal
* Taking Chromium Supplement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Every patient; who is over/and 18 years old age, admitted to Anesthesiology Intensive Care Unit, agreed to participate in the study (with informed consent) and not - taking chromium supplement
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss this matter with all the researchers and ethics committee.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were admitted to the anesthesiology intensive care unit and met the inclusion criteria were recruited between February 2024 and August 2024. The first participant was enrolled on February 7, 2024, and the last participant was enrolled, and primary outcome data collection was completed on August 8, 2024. The study was fully completed on August 14, 2024, following the collection of all secondary outcomes.
Pre-assignment Details: All of the enrolled participants were included in the study.
Groups:
- Intensive Care Patients: Patients who are admitted to the intensive care unit.
Period: Overall Study
Arm/Group | Intensive Care Patients
Started | 309
Completed | 309
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.72 (16.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167
  Male | 142
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: Centimeters] | 165.21 (9.03)
Body Mass [Mean (Standard Deviation); unit: Kilograms] | 73.8 (15.81)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27 (5.36)
Comorbidities [Number; unit: participants]
  Cardiovascular Diseases | 202
  Diabetes | 89
  Malignancy | 79
  Neurological Disorders | 76
  Respiratory Diseases | 69
  Liver Diseases | 4
Reason for Intensive Care Admission [Count of Participants; unit: Participants]
  Postoperative Care | 216
  Respiratory Distress | 45
  Sepsis | 31
  Neurological Disorders | 10
  Trauma | 5
  Drug Intoxication | 2
SOFA Score [Mean (Standard Deviation); unit: Scores on a scale] — The Sequential Organ Failure Assessment (SOFA) score is a simple method of assessing and monitoring organ dysfunction in critically ill patients. Each organ system (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) receives a score ranging from 0 (normal) to 4 (most abnormal), with a minimum SOFA score of 0 and a maximum SOFA score of 24. The higher the SOFA score, the higher the likely mortality.
  Scores on a scale | 0.91 (1.77)
APACHE - II Score [Mean (Standard Deviation); unit: Scores on a scale] — Acute Physiology and Chronic Health Evaluation - II (APACHE - II) score is a general measure of disease severity based on current physiologic measurements (body temperature, heart and respiratory rate, mean arterial pressure, pH), age & previous health conditions. The score can help in the assessment of patients to determine the level and degree of diagnostic and therapeutic intervention. The range of APACHE - II score is 0 (minimum) to 71 (maximum); increasing score is associated with an increasing risk of hospital death.
  Scores on a scale | 9.33 (5.65)
Nutritional Status [Count of Participants; unit: Participants] — Nutritional statuses of patients were recorded to examine its effects on serum chromium levels and also, mortality.
  Participants
    Enteral | 265
    Parenteral | 2
    Enteral and Parenteral | 42

OUTCOME MEASURES:

1. Primary Outcome: Serum Chromium Level
Description: Serum chromium levels of participants were measured once a week throughout the participant's ICU stay, starting from admission. The healthy reference range of 0.7 to 28.0 µg/L for blood chromium levels was used.
Time Frame: Once a week throughout the participant's ICU stay, starting from admission (day 0, day 7, day 14 and day 21).
Population: A total of 309 participants were included in the study. Measurements were taken once a week throughout their hospital stay. In the first measurement (ICU admission/day 0), 309 participants; in the second measurement (participants who completed the 7th day of ICU stay), 51 participants; in the third measurement (participants who completed the 14th day of ICU stay), 24 participants; and in the fourth measurement (participants who completed the 21st day of ICU stay), 13 participants were assessed.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 309
µg/L
  First Measurement (Day 0) | 8.93 (5.18)
  Second Measurement (Day 7): number analyzed (Participants) | 51
  Second Measurement (Day 7) | 9.74 (5.31)
  Third Measurement (Day 14): number analyzed (Participants) | 24
  Third Measurement (Day 14) | 9.68 (4.41)
  Fourth Measurement (Day 21): number analyzed (Participants) | 13
  Fourth Measurement (Day 21) | 11.01 (4.03)

2. Secondary Outcome: HbA1c
Description: The HbA1c level when the participant is admitted to the intensive care unit. Possible levels are less/equal/more than %6,5.
Time Frame: At the time of ICU admission (day 0).
Measure: Mean (Standard Deviation); unit: Percentage of glycated hemoglobin (%)
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 309
Percentage of glycated hemoglobin (%) | 5.99 (1.04)

3. Secondary Outcome: Blood Glucose
Description: During the ICU stay, participants underwent daily blood glucose measurements using the fingertip method. Weekly averages of the measurements were calculated. Although there is no accepted definition of acute hyperglycemia in the critical care setting, it is generally considered to be above 180 - 220 mg/dL. In our study, we considered the value of 200 mg/dL as a threshold for stress hyperglycemia.
Time Frame: Week 1, week 2, week 3 and week 4.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 309
mg/dL
  First Measurement (Week 1) | 128.68 (35.97)
  Second Measurement (Week 2) | 122.25 (27.43)
  Third Measurement (Week 3) | 122.29 (24.47)
  Fourth Measurement (Week 4) | 116.46 (30.8)

4. Secondary Outcome: Lipid Profile
Description: Lipid Profiles (HDL, LDL, Triglycerides, Total Cholesterol) of participants were measured once a week throughout the participant's ICU stay, starting from admission. The optimal lipid levels vary depending on age, gender, and other risk factors; however, they are generally recommended within the following ranges:
  * LDL cholesterol: Less than 100 mg/dL,
  * HDL cholesterol: Greater than 40 mg/dL for men and greater than 50 mg/dL for women,
  * Triglycerides: Less than 150 mg/dL,
  * Total cholesterol: Less than 200 mg/dL.
Time Frame: Once a week throughout the participant's ICU stay, starting from admission (day 0, day 7, day 14 and day 21).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 309
mg/dL
  First Triglycerides Measurement (Day 0) | 118.28 (74.21)
  Second Triglycerides Measurement (Day 7): number analyzed (Participants) | 51
  Second Triglycerides Measurement (Day 7) | 135.06 (58.83)
  Third Triglycerides Measurement (Day 14): number analyzed (Participants) | 24
  Third Triglycerides Measurement (Day 14) | 124.29 (57.62)
  Fourth Triglycerides Measurement (Day 21): number analyzed (Participants) | 13
  Fourth Triglycerides Measurement (Day 21) | 145.23 (81.89)
  First HDL Measurement (Day 0) | 38.93 (12.08)
  Second HDL Measurement (Day 7): number analyzed (Participants) | 51
  Second HDL Measurement (Day 7) | 29.7 (11.92)
  Third HDL Measurement (Day 14): number analyzed (Participants) | 24
  Third HDL Measurement (Day 14) | 23.9 (12.63)
  Fourth HDL Measurement (Day 21): number analyzed (Participants) | 13
  Fourth HDL Measurement (Day 21) | 22.84 (11.01)
  First LDL Measurement (Day 0) | 92.34 (34.64)
  Second LDL Measurement (Day 7): number analyzed (Participants) | 51
  Second LDL Measurement (Day 7) | 75.1 (35.28)
  Third LDL Measurement (Day 14): number analyzed (Participants) | 24
  Third LDL Measurement (Day 14) | 57.51 (37.25)
  Fourth LDL Measurement (Day 21): number analyzed (Participants) | 13
  Fourth LDL Measurement (Day 21) | 57.69 (26.51)
  First VLDL Measurement (Day 0) | 23.86 (14.85)
  Second VLDL Measurement (Day 7): number analyzed (Participants) | 51
  Second VLDL Measurement (Day 7) | 26.73 (12.29)
  Third VLDL Measurement (Day 14): number analyzed (Participants) | 24
  Third VLDL Measurement (Day 14) | 24.77 (11.64)
  Fourth VLDL Measurement (Day 21): number analyzed (Participants) | 13
  Fourth VLDL Measurement (Day 21) | 31.31 (23.04)
  First Total Cholesterol Measurement (Day 0) | 143.14 (45.79)
  Second Total Cholesterol Measurement (Day 7): number analyzed (Participants) | 51
  Second Total Cholesterol Measurement (Day 7) | 116.14 (46.59)
  Third Total Cholesterol Measurement (Day 14): number analyzed (Participants) | 24
  Third Total Cholesterol Measurement (Day 14) | 89.25 (55.01)
  Fourth Total Cholesterol Measurement (Day 21): number analyzed (Participants) | 13
  Fourth Total Cholesterol Measurement (Day 21) | 82.92 (42.03)

5. Secondary Outcome: Glycemic Variability - Coefficient of Variation (CV)
Description: The coefficient of variation (CV) is the standard deviation divided by the mean of the glycemic values. A higher coefficient of variation is associated with greater glycemic variability. A CV of < 36% is a good threshold. The coefficients of variation were calculated after each participant was discharged from the ICU, based on all the blood glucose values measured during their stay.
Time Frame: During each participant's ICU stay (ranging from 1 to 4 weeks).
Measure: Mean (Standard Deviation); unit: Percentage of coefficient of variation
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 309
Percentage of coefficient of variation | 22.01 (12.24)

ADVERSE EVENTS:
Time Frame: All - cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Description: All - cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Arm/Group | Intensive Care Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT06334042/Prot_SAP_000.pdf